CLINICAL TRIAL: NCT00028938
Title: A Phase III Randomized Trial Evaluating the Effect of Epoetin Alfa (Procrit) on Local Control in Patients Undergoing Concurrent Chemotherapy and Radiation Therapy for Non-Small Cell Lung Cancer
Brief Title: Chemotherapy and Radiation Therapy With or Without Epoetin Alfa in Treating Patients With Stage IIIA or Stage IIIB Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: REBACDR0000069148; CCCWFU-62299; CCCWFU-BG01-193; NCI-P01-0200
Record Dates: First submitted 2002-01-04; First posted 2003-07-01 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Lung Cancer
Keywords: squamous cell lung cancer; large cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Epoetin Alfa; Carboplatin; Paclitaxel; Radiotherapy

INTERVENTIONS:
Biological: epoetin alfa
Drug: carboplatin
Drug: paclitaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Epoetin alfa may stimulate red blood cell production and prevent or treat anemia in patients who are undergoing radiation therapy and chemotherapy. It is not yet known if chemotherapy combined with radiation therapy is more effective with or without epoetin alfa in treating non-small cell lung cancer.

PURPOSE: Randomized phase III trial to determine the effectiveness of chemotherapy combined with radiation therapy with or without epoetin alfa in treating patients who have stage IIIA or stage IIIB non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of epoetin alfa in maintaining hemoglobin levels in patients with stage IIIA or IIIB non-small cell lung cancer when treated with chemoradiotherapy.
* Compare the time to local and systemic progression in patients receiving chemoradiotherapy with or without epoetin alfa.
* Compare tumor response rate and overall survival in patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare quality of life in patients treated with these regimens.
* Compare the number of transfusions in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to Karnofsky performance status (90-100% vs 60-80%), weight loss (no more than 5% vs 6-10%), and baseline hemoglobin (women 11.0-12.4 g/dL and men 11.0-13.4 g/dL vs women 12.5-15.0 g/dL and men 13.5-15.0 g/dL). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Beginning 7-10 days before the start of chemoradiotherapy, patients receive epoetin alfa subcutaneously once weekly for 8 weeks. Patients receive paclitaxel IV over 1 hour and carboplatin IV over 30 minutes once weekly for 7 weeks. Patients undergo radiotherapy 5 days a week for 7 weeks for a total of 33 treatments. Treatment continues in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive paclitaxel, carboplatin, and radiotherapy as in arm I. Quality of life is assessed at baseline, at completion of chemoradiotherapy, every 3 months for 1 year, every 4 months for 1 year, and then every 6 months for 3 years.

Patients are followed every 3 months for 1 year, every 4 months for 1 year, and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 202-232 patients (101-116 per treatment arm) will be accrued for this study within 1.7-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage IIIA or IIIB non-small cell lung cancer (NSCLC)

  * Squamous cell carcinoma
  * Adenocarcinoma (including bronchoalveolar cell)
  * Large cell anaplastic carcinoma (including giant and clear cell carcinomas)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin 11.0-15 g/dL
* If hemoglobin is 11.0-11.9 g/dL then the following lab values are required:

  * Iron greater than 60 mcg/mL
  * Transferrin saturation greater than 20%
  * Ferritin at least 100 mg/mL
  * Iron binding capacity less than 400 mcg/dL
  * RBC folate normal
  * B12 normal

Hepatic:

* Bilirubin less than 1.5 mg/dL
* AST less than 2 times upper limit of normal

Renal:

* Creatinine clearance at least 20 mL/min

Cardiovascular:

* No uncontrolled hypertension

Pulmonary:

* FEV1 at least 0.8 L

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known hypersensitivity to mammalian cell-derived products or human albumin
* No other concurrent or prior malignancy within the past 2 years except non- melanoma skin cancers

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 30 days since prior transfusion
* No prior epoetin alfa or experimental forms of epoetin alfa

Chemotherapy:

* No prior chemotherapy for NSCLC

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy for NSCLC

Surgery:

* At least 2 weeks since prior thoracotomy

Other:

* No concurrent therapy for iron, folate, or B12 deficiency
* No other concurrent anti-cancer therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2002-01-01 (Actual); Primary Completion 2002-11-10 (Actual); Study Completion 2002-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur William Blackstock, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina, United States